CLINICAL TRIAL: NCT06405997
Title: The Genotype and Phenotype of Lymphangioleiomyomatosis
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202401140RINE
Record Dates: First submitted 2024-05-02; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-04

CONDITIONS: Sporadic Lymphangioleiomyomatosis; TSC-associated Lymphangioleiomyomatosis
Keywords: Lymphangioleiomyomatosis
MeSH Terms: conditions — Lymphangioleiomyomatosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to differentiate between sporadic Lymphangioleiomyomatosis and Tuberous Sclerosis Complex-associated Lymphangioleiomyomatosis.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 y/o
* Patient with Chest CT showed cystic lung disease, suspected Lymphangioleiomyomatosis

Exclusion Criteria:

* age < 18 y/o

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Chest CT showed cystic lung disease, suspected Lymphangioleiomyomatosis in National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-05-10 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
The genotype and phenotype of lymphangioleiomyomatosis | one month

CONTACTS AND LOCATIONS:
Overall Officials: Yao-Wen Kuo, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan